CLINICAL TRIAL: NCT04180605
Title: The Value of FEops HEARTguideTM Patient-Specific Computational Simulation in the Planning of Percutaneous Left Atrial Appendage Closure With the AmplatzerTM AmuletTM Device (PREDICT-LAA)
Brief Title: Computational Simulation to Plan for Percutaneous Left Atrial Appendage Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Feops (Industry); Abbott (Industry)
Responsible Party: Principal Investigator, Ole De Backer, Dr. Ole De Backer, MD, PhD, Consultant Interventional Cardiology, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-19043746 - PREDICT-LAA
Record Dates: First submitted 2019-11-21; First posted 2019-11-27 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation; Stroke Prevention
Keywords: Atrial fibrillation; Left atrial appendage; Transcatheter closure; Stroke prevention; Computed tomography; Computational simulation; Preoperative planning
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Intervention Model Description: 200 patients selected for percutaneous LAA closure with an AmplatzerTM AmuletTM device will be enrolled in this study and randomized into the following two arms: the comparator (standard of care arm) for whom the procedure will be conducted following the standard of care of the center, and the computational simulation arm where the pre-procedural planning will include a careful analysis of the computational simulation results provided by the FEops HEARTguideTM platform.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care treatment arm (Active Comparator): When patients are randomized to the standard treatment arm, patients will be treated according to the participating site's routine practice. As pre-procedural imaging, a cardiac CT-scan has to be performed; this can also be complemented with TEE at the discretion of the operator. The LAA closure procedure should be performed according to routine practice of the participating site - either in general or local anesthesia.
  For those cases randomized to the standard treatment arm, the pre-procedural CT-scans will still be collected at completion of the study and FEops HEARTguideTM simulations will be generated, blinded for the procedural images and outcome. These simulations will be compared with the final device size and implant position and will be used for an additional comparative PREDICT-LAA sub-study.
  Interventions: Procedure: Left atrial appendage closure
- Computational simulation arm (Experimental): When patients are randomized to the computational simulation arm, the procedure will still be performed according to the participating site's routine practice - however, the procedure will only be performed after careful review of the FEops HEARTguideTM simulation results. The only prerequisite is that all patients randomized to this arm will have to undergo a pre-procedural cardiac CT-scan that will be uploaded into the FEops HEARTguideTM platform. Following this upload, a pre-procedural simulation plan will be provided to the operator, containing a set of optimal and suboptimal closure device sizes and implant positions. Software and technology upgrades of the FEops HEARTguideTM platform will be allowed during the course of the study.
  Interventions: Other: Additional support for preoperative planning of LAA closure procedures; Procedure: Left atrial appendage closure

INTERVENTIONS:
Other: Additional support for preoperative planning of LAA closure procedures — The results of the computational simulations provided by FEops HEARTguideTM will be used in the "computational simulation arm" as an additional preoperative planning tool and their potential added value will be assessed by comparison to the standard of care arm.
  Arms: Computational simulation arm
Procedure: Left atrial appendage closure — Transcatheter device insertion to exclude the LAA from the cardiac circulation

SUMMARY:
To ensure a successful percutaneous left atrial appendage (LAA) closure, it is important to select the correct size of the closure device used for each patient. To define and measure the size of the LAA, 2D transesophageal echocardiography (TEE) has been typically used. An increasing number of hospitals recently switched to measure the size of the LAA using a cardiac computed tomography (CT) scan. Although this CT scan helps to better define and measure the LAA, it is still difficult to determine the exact anticipated 'landing zone' or 'position' of the closure device. A novel strategy of preprocedural planning includes the use of preoperative computer simulations based on CT imaging (Feops HEARTguideTM), where the device is deployed with a computer simulation into the patient-specific LAA anatomy to provide the operator both optimal and suboptimal scenario's showing different sizes and positions of the closure device.

The aim of this study is to assess whether use of FEops HEARTguide computer simulations based on cardiac CT-imaging can contribute to a better preprocedural planning and improved procedural outcomes of percutaneous LAA closure procedures with an Amplatzer Amulet device.

The PREDICT-LAA trial will investigate the possible positive effect of a computer simulation using a CT scan of the LAA performed prior to the procedure. The hypothesis is that by using this new computer simulation, better planning of the intervention can be obtained.

DETAILED DESCRIPTION:
To prevent stroke in patients with non-valvular atrial fibrillation (NVAF) and contraindication(s) to oral anticoagulant therapy, percutaneous left atrial appendage (LAA) closure is increasily being chosen as an alternative therapeutic option. To obtain a successful percutaneous LAA closure, an accurate preoperative planning is required to understand the LAA morphology and assess the correct size and optimal position of the device. The instructions for use (IFUs) of the medical device providers are still based on two-dimensional transesophageal echocardiography, whereas an increasing number of centers have shifted towards LAA sizing and planning based on cardiac computed tomography (CT) images. Other options are also available for preoperative planning, among others the use of 3D printed LAA models. However, this has a number of disadvantages, among others complex logistics and the possible inaccuracy in terms of mechanical response of the printing material used for the 3D printed model.

Based on the FEops HEARTguideTM platform, a computational model for percutaneous LAA closure was developed and validated. The computer simulations are based on CT images, and can predict different possible LAA closure options for the patient, including optimal and suboptimal sizing and positioning of the LAA closure device. This can be achieved by modelling the mechanical interaction between the device and the 3D patient-specific LAA anatomy reconstructed from the CT images. The results are available as a web-based 3D-viewer and allow the physician to analyse the different device size and implant position options prior to the procedure.

The PREDICT-LAA trial aims to study the possible added value of FEops HEARTguideTM patient-specific computational simulation in the planning of percutaneous LAA closure with the AmplatzerTM AmuletTM device, with special focus on procedural safety and efficiency as well as on clinical outcomes.

The PREDICT-LAA study is a prospective, multicenter, randomized controlled trial. In total, 200 patients eligible for percutaneous LAA closure with an AmplatzerTM AmuletTM device (Abbott, USA) will be enrolled - 100 patients will be allocated to the computational simulation treatment arm and 100 patients to the standard treatment arm.

All participants will be treated according to the standard of care of the center - additionally, the preoperative planning for patients allocated to the computational simulation treatment arm will include a careful analysis of the computational simulation results provided by the FEops HEARTguideTM platform.

Patients with non-valvular atrial fibrillation who are referred to and deemed eligible for percutaneous LAA closure with an AmplatzerTM AmuletTM closure device can be included. Patients with reduced renal function, known contrast agent allergy, and/or suboptimal cardiac CT-image quality are excluded from this trial.

The participant shall be informed about the aim and procedure of the PREDICT-LAA study and written informed consent shall be obtained in order to include the participant.

All patients enrolled in the PREDICT-LAA study should have a post-procedural cardiac CT scan at three months after the LAA closure procedure to check for complete LAA closure, device-related thrombosis (DRT) and device position. The CT CoreLab for assessment of this post-procedural CT-scans will be performed at Rigshospitalet, Copenhagen, Denmark. The readers of the CT-scan will be blinded from the baseline data, randomisation arm and procedural data.

The risk related to this study and, in particular, the CT-scan is low - especially as patients with renal insufficiency, iodine contrast allergy and/or contraindications for CT-scan are excluded. Concerning the radiation dose of maximally two CT-scans, we can report that patients will receive a radiation dose of 6 to 15 mSievert, depending on weight and heart frequency/rhythym. It can be calculated that lifetime risk to die from cancer, hereby, theoretically increases with maximally 0,06%. Thus, the patients' lifetime risk to die from cancer increases from 25.0% to 25.06%.

The patients are informed about the aim and procedure of the study and are only included in case of written consent. Unknown side effects or risks associated with the study cannot be ruled-out.

The protocol of the trial has been approved by local regional Ethics Committees in each participating country, the collection of data complies with the regulatory rules of the Danish Data Protection Agency, and the study is being conducted in compliance with good clinical practice and with the Helsinki II Declaration as adopted by the 18th World Medical Assembly in Helsinki, Finland, in 1964 and subsequent versions.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Patients with non-valvular atrial fibrillation (NVAF) who are referred to and approved for percutaneous LAA closure with an Amplatzer Amulet closure device, according to local practice and legislation.
* Written informed consent.

Exclusion Criteria:

* Reduced renal function with eGFR < 30 mL/min/1.73 m^2.
* Iodine contrast allergy or other condition that prohibits cardiac CT imaging.
* Suboptimal image quality of the pre-procedural cardiac CT-scan.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incomplete LAA closure and definite device-related thrombosis (DRT) | Post-procedural cardiac CT scan at 3 months after LAA closure
  The percentage of patients with incomplete LAA closure (defined as any remaining contrast leakage into the LAA distal of the Amulet lobe) and/or a definite DRT at post-procedural cardiac CT imaging at three months after the procedure. Definite DRT is defined as "high-grade" hypo-attenuating thickening at the atrial surface of the closure device - as previously described by Korsholm et al., Circ Cardiovasc Interv, 2019.

SECONDARY OUTCOMES:
Number of closure devices used | Periprocedural
  Number of LAA closure devices used per procedure
Number of repositioning | Periprocedural
  Number of LAA closure device repositionings per procedure. Repositioning is defined as full deployment of the Amulet lobe in the LAA, followed by either a full or partial recapture and re-deployment of the Amulet lobe
Procedural time | Periprocedural
  Duration of the LAA closure procedure [minutes]
Radiation exposure | Periprocedural
  Radiation exposure per procedure [Gy]
Contrast medium | Periprocedural
  Amount of contrast medium used per procedure [mL]
Procedural-related complications | Periprocedural and between randomization and within 7 days of the procedure
  Recording of the following events if any:
  * LAA closure device embolization
  * Pericardial effusion requiring intervention
  * Procedure-related stroke
  * Procedure-related death
Final position of the device | During post-procedural cardiac CT scan at 3 months after LAA closure
  Coverage of all LAA trabeculations by the Amulet shaped disc of the Amulet lobe/disc and a concave device without retraction of the disc into the LAA
Composite of all-cause death and thromboembolic event | 12 months after randomization
  Recording of the following events if any: transient ischemic attack, ischemic stroke, systemic embolism
Different degrees of contrast leakage into the LAA | Post-procedural cardiac CT scan at 3 months after LAA closure
  Different degrees of contrast leakage into the LAA

CONTACTS AND LOCATIONS:
Overall Officials: Ole De Backer, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (12):
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Hopital Civil Marie Curie CHU de Charleroi, Charleroi
- Canada (2):
  - Montreal Heart Institute, Montreal
  - Vancouver General Hospital, Vancouver
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (2):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Institut Cardiovasculaire Paris Sud, Massy
- Fondazione Toscana G. Monasterio, Massa, Italy
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Background] Chow DH, Bieliauskas G, Sawaya FJ, Millan-Iturbe O, Kofoed KF, Sondergaard L, De Backer O. A comparative study of different imaging modalities for successful percutaneous left atrial appendage closure. Open Heart. 2017 Jun 30;4(2):e000627. doi: 10.1136/openhrt-2017-000627. eCollection 2017. PMID 28761682
- [Background] Korsholm K, Jensen JM, Nielsen-Kudsk JE. Intracardiac Echocardiography From the Left Atrium for Procedural Guidance of Transcatheter Left Atrial Appendage Occlusion. JACC Cardiovasc Interv. 2017 Nov 13;10(21):2198-2206. doi: 10.1016/j.jcin.2017.06.057. Epub 2017 Aug 30. PMID 28866042
- [Background] Otton JM, Spina R, Sulas R, Subbiah RN, Jacobs N, Muller DW, Gunalingam B. Left Atrial Appendage Closure Guided by Personalized 3D-Printed Cardiac Reconstruction. JACC Cardiovasc Interv. 2015 Jun;8(7):1004-6. doi: 10.1016/j.jcin.2015.03.015. No abstract available. PMID 26088522
- [Background] de Jaegere P, Rocatello G, Prendergast BD, de Backer O, Van Mieghem NM, Rajani R. Patient-specific computer simulation for transcatheter cardiac interventions: what a clinician needs to know. Heart. 2019 Mar;105(Suppl 2):s21-s27. doi: 10.1136/heartjnl-2018-313514. PMID 30846521
- [Background] Rocatello G, El Faquir N, De Santis G, Iannaccone F, Bosmans J, De Backer O, Sondergaard L, Segers P, De Beule M, de Jaegere P, Mortier P. Patient-Specific Computer Simulation to Elucidate the Role of Contact Pressure in the Development of New Conduction Abnormalities After Catheter-Based Implantation of a Self-Expanding Aortic Valve. Circ Cardiovasc Interv. 2018 Feb;11(2):e005344. doi: 10.1161/CIRCINTERVENTIONS.117.005344. PMID 29386188
- [Background] Bavo AM, Wilkins BT, Garot P, De Bock S, Saw J, Sondergaard L, De Backer O, Iannaccone F. Validation of a computational model aiming to optimize preprocedural planning in percutaneous left atrial appendage closure. J Cardiovasc Comput Tomogr. 2020 Mar-Apr;14(2):149-154. doi: 10.1016/j.jcct.2019.08.010. Epub 2019 Aug 20. PMID 31445885
- [Derived] De Backer O, Iriart X, Kefer J, Nielsen-Kudsk JE, Aminian A, Rosseel L, Kofoed KF, Odenstedt J, Berti S, Saw J, Sondergaard L, Garot P. Impact of Computational Modeling on Transcatheter Left Atrial Appendage Closure Efficiency and Outcomes. JACC Cardiovasc Interv. 2023 Mar 27;16(6):655-666. doi: 10.1016/j.jcin.2023.01.008. Epub 2023 Feb 22. PMID 36990554
- [Derived] Swaans MJ, Huijboom MFM, Boersma LVA. Fluoroscopic Guidance: An Echo From the Past? JACC Cardiovasc Interv. 2021 Aug 23;14(16):1827-1829. doi: 10.1016/j.jcin.2021.07.003. No abstract available. PMID 34412800
- [Derived] Garot P, Iriart X, Aminian A, Kefer J, Freixa X, Cruz-Gonzalez I, Berti S, Rosseel L, Ibrahim R, Korsholm K, Odenstedt J, Nielsen-Kudsk JE, Saw J, Sondergaard L, De Backer O. Value of FEops HEARTguide patient-specific computational simulations in the planning of left atrial appendage closure with the Amplatzer Amulet closure device: rationale and design of the PREDICT-LAA study. Open Heart. 2020 Aug;7(2):e001326. doi: 10.1136/openhrt-2020-001326. PMID 32763967